CLINICAL TRIAL: NCT05320172
Title: Effect of Platelet Rich Plasma Eye Drops in Corneal Surface Diseases
Brief Title: Platelet Rich Plasma in Corneal Surface Diseases
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelnasser Mohamed Abdelnasser, Ophthalmology Resident, Assiut University Hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP ED in corneal diseases
Record Dates: First submitted 2021-11-16; First posted 2022-04-11 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Persistent Corneal Epithelial Defects; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Fifty milliliters of whole blood will be placed in five 10-ml vacutainer tubes containing anticoagulant-citrate-dextrose solution (1.4 ml) and centrifuged at 200g for 11 min. The upper two layers of the centrifuged blood, the plasma and buffy coat layer will be separated in a sterile manner and diluted to 20 % (v/v) with a sterile saline solution. The final preparation is divided into 5-ml bottles wrapped in aluminum foil for protection from ultraviolet light. The patients are instructed to store these bottles at -20 °C until required. The bottles being used will be maintained under refrigerated conditions at 4 °C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Participants with persistent epithelial defects will be treated with autologous platelet rich plasma eye drops.
  Interventions: Drug: Autologous platelet rich plasma eye drops

INTERVENTIONS:
Drug: Autologous platelet rich plasma eye drops — Fifty milliliters of patient's own whole blood will be placed in five 10-ml vacutainer tubes containing anticoagulant-citrate-dextrose solution (1.4 ml) and centrifuged at 200g for 11 min. The upper two layers of the centrifuged blood, the plasma and buffy coat layer will be separated in a sterile manner and diluted to 20 % (v/v) with a sterile saline solution. The final preparation is divided into 5-ml bottles wrapped in aluminum foil for protection from ultraviolet light. The patients are instructed to store these bottles at -20 °C until required. The bottles being used will be maintained under refrigerated conditions at 4 °C.
  Other Names: PRP eye drops

SUMMARY:
The Aim of the study is to evaluate the efficacy of platelet rich plasma eye drops in the management of different corneal surface disorders.

PRP is a blood sample with a concentrated platelet count, and numerous growth factors that are associated with conjunctival and corneal wound healing process. which is an important advantage over other products. PRP eye drops recently are proving to be an effective and potent therapeutic approach to promote corneal wound re-epithelization and promote ocular surface regeneration in different pathological conditions.

DETAILED DESCRIPTION:
There are many conditions in which the ocular surface is severely affected as keratoconjunctivitis sicca, persistent epithelial corneal defect, recurrent corneal erosion, neurotrophic keratopathy, post laser in-situ keratomileusis (LASIK) ocular surface syndrome (OSS), dormant corneal ulcer, graft-versus-host disease, ocular cicatricial pemphigoid, and neurotrophic changes. If corneal wound healing does not occur promptly, it can lead to visual loss, severe scarring, infection and even corneal perforation, the treatment of ocular surface disorders has a multifactorial approach and conventional therapy is often not enough to solve the problem.

Platelet-rich plasma (PRP) is defined as a portion of the plasma fraction of autologous blood having a platelet concentration above baseline. They use a PRP device, concentrate platelets using a double centrifugation technique and activate PRP just when they are ready to use it. The final concentration is at least 1.000.000 platelets/ microliter. Therefore, it is an autologous concentration of platelets and growth factors.

An important reservoir of proteins and growth factors precipitating in haemostasis, tissue regeneration, immune response, and wound healing. Alpha granules of the platelets include over 30 biologically active substances such as platelet-derived growth factor, transforming growth factor b1 and b2 and insulin-like growth factor 1, vascular endothelial growth factor, epidermal cell growth factor, fibroblast growth factor 2, and insulin-like growth factor.

Eye platelet-rich plasma has a lubricating effect and has been effective in regenerating the ocular surface in cases of micropunctate keratitis, decreasing inflammation in patients suffering from dry eye and stimulating wound-healing processes in dormant corneal ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent epithelial defects (Exposure keratopathy, Post infectious keratitis).
2. Dry eye disease.

Exclusion Criteria:

1. Active ocular infection or inflammation.
2. Patients will be withdrawn if allergic or adverse side effects develop.
3. Pregnancy or breast feeding.
4. The use of systemic antiplatelet or anticoagulant.
5. Uncontrolled systemic diseases
6. Non-compliance with the study protocol.
7. Positive HIV, HBV, HCB or Syphilis.
8. Anemia (less than 10 g/dl of HGB, platelet count less than 105/ul).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of platelet rich plasma eye drops in the management of persistent corneal epithelial defects, and dry eye disease by observation of change in size of defect over different periods of time. | At 48 hours, one week and one month.
  To evaluate the effect of platelet-rich plasma (PRP) eye drops in management of different ocular surface pathologies, the therapeutic response will be evaluated with clinical examination and follow up.
  Main outcome measurements include the change in size of defect by fluorescein staining on slit lamp biomicroscopy.
  The largest linear dimension of the epithelial defect and its largest possible perpendicular within the confines of the epithelial defect are measured in millimeters using a slit lamp.
Evaluation of the efficacy of platelet rich plasma eye drops in the management of persistent corneal epithelial defects, and dry eye disease by observation of change in visual acuity. | At 48 hours, one week and one month.
  To evaluate the effect of platelet-rich plasma (PRP) eye drops in management of different ocular surface pathologies, the therapeutic response will be evaluated with clinical examination and follow up.
  Main outcome measurements include the change in visual acuity measured by Snellen visual acuity (VA) testing.
Evaluation of the efficacy of platelet rich plasma eye drops in the management of persistent corneal epithelial defects, and dry eye disease by observation of change in height of tear meniscus, | At 48 hours, one week and one month.
  To evaluate the effect of platelet-rich plasma (PRP) eye drops in management of different ocular surface pathologies, the therapeutic response will be evaluated with clinical examination and follow up.
  Main outcome measurements include the change in height of tear meniscus measured by slit lamp biomicroscopy.

SECONDARY OUTCOMES:
Evaluation of the efficacy of platelet rich plasma eye drops in the relief symptoms caused by persistent corneal epithelial defects, and dry eye disease by observation of change in ocular symptoms. | At 48 hours, one week and one month.
  Secondary outcome measurements include the change and improvement of subjective symptoms during treatment; particularly pain. assessed by visual analog score for pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Abdelrahman, MD, Study Chair — Professor of ophthalmology, Faculty of medicine, Assiut University; Mahmoud F Rateb, MD, Study Chair — Assistant professor of ophthalmology, Faculty of medicine, Assiut University; Mohamed G Saleh, MD, Study Director — Lecturer of ophthalmology, Faculty of medicine, Assiut university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim KM, Shin YT, Kim HK. Effect of autologous platelet-rich plasma on persistent corneal epithelial defect after infectious keratitis. Jpn J Ophthalmol. 2012 Nov;56(6):544-50. doi: 10.1007/s10384-012-0175-y. Epub 2012 Sep 13. PMID 22972393
- [Result] Noble BA, Loh RS, MacLennan S, Pesudovs K, Reynolds A, Bridges LR, Burr J, Stewart O, Quereshi S. Comparison of autologous serum eye drops with conventional therapy in a randomised controlled crossover trial for ocular surface disease. Br J Ophthalmol. 2004 May;88(5):647-52. doi: 10.1136/bjo.2003.026211. PMID 15090417
- [Result] Alio JL, Arnalich-Montiel F, Rodriguez AE. The role of "eye platelet rich plasma" (E-PRP) for wound healing in ophthalmology. Curr Pharm Biotechnol. 2012 Jun;13(7):1257-65. doi: 10.2174/138920112800624355. PMID 21740369
- [Result] Alio JL, Abad M, Artola A, Rodriguez-Prats JL, Pastor S, Ruiz-Colecha J. Use of autologous platelet-rich plasma in the treatment of dormant corneal ulcers. Ophthalmology. 2007 Jul;114(7):1286-1293.e1. doi: 10.1016/j.ophtha.2006.10.044. Epub 2007 Feb 26. PMID 17324465
- [Result] Nurden AT. Platelets, inflammation and tissue regeneration. Thromb Haemost. 2011 May;105 Suppl 1:S13-33. doi: 10.1160/THS10-11-0720. Epub 2011 Apr 11. PMID 21479340
- [Result] Lee JH, Kim MJ, Ha SW, Kim HK. Autologous Platelet-rich Plasma Eye Drops in the Treatment of Recurrent Corneal Erosions. Korean J Ophthalmol. 2016 Apr;30(2):101-7. doi: 10.3341/kjo.2016.30.2.101. Epub 2016 Mar 25. PMID 27051257
- [Result] Wu TE, Chen CJ, Hu CC, Cheng CK. Easy-to-prepare autologous platelet-rich plasma in the treatment of refractory corneal ulcers. Taiwan J Ophthalmol. 2015 Jul-Sep;5(3):132-135. doi: 10.1016/j.tjo.2014.09.001. Epub 2014 Nov 20. PMID 29018685
- See also: Eye platelet-rich plasma in the treatment of ocular surface disorders — https://www.ophed.com/system/files/2015/07/Eye%20platelet-rich%20plasma%20in%20the%20treatment%20of%20ocular%20surface%20disorders.pdf?fbclid=IwAR3A7EUT-g_PraOMio5VqndyDA0i5h1SRQa35gKFtP7r4xqvX1hxr1YrP1g
- See also: Platelet-Rich Plasma (PRP): What Is PRP and What Is Not PRP? Marx, Robert E. DDS — https://journals.lww.com/implantdent/Fulltext/2001/10000/Platelet_Rich_Plasma__PRP___What_Is_PRP_and_What.2.aspx
- See also: Treatment of Dry Eye Disease with Autologous Platelet-Rich Plasma — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5693817/